CLINICAL TRIAL: NCT05672420
Title: A Multicenter, Phase Ib/II Trial of the Safety and Efficacy of Umbilical Cord Derived Mesenchymal Stem Cells in Treatment-induced Myelosuppression in Patients With Hematologic Malignancies (USMYE Trial)
Brief Title: Umbilical Cord Derived Mesenchymal Stem Cells for Treatment-induced Myelosuppression in Hematologic Malignancies
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Collaborators: Wuhan TongJi Hospital (Other); Wuhan Central Hospital (Other)
Responsible Party: Principal Investigator, Qiubai Li, M.D. & Ph.D., Professor, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UHCT22668
Record Dates: First submitted 2023-01-01; First posted 2023-01-05 (Actual); Last update posted 2023-01-05 (Actual); Status verified 2023-01

CONDITIONS: Hematologic Neoplasms; Neutropenia; Anemia; Thrombocytopenia; Infections; Bleeding
Keywords: umbilical cord derived mesenchymal stem cells; treatment-induced myelosuppression; neutropenia; anemia; thrombocytopenia; infections; bleeding; hematologic malignancies; leukemia; lymphoma; multiple myeloma; chemotherapy; targeted therapy; hematopoietic stem cell transplantation
MeSH Terms: conditions — Hematologic Neoplasms; Neutropenia; Anemia; Thrombocytopenia; Infections; Hemorrhage; Leukemia; Lymphoma; Multiple Myeloma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- umbilical cord derived mesenchymal stem cells (UC-MSCs) (Experimental): In the Phase Ib study, participants will be those with treatment-induced myelosuppression and acute myeloid leukemia/acute lymphoblastic leukemia, UC-MSCs will be preset with 5 escalation dose levels: dose A , dose B, dose C ,dose D and dose E, frequency of infusion will be preset with 3 escalation levels: frequency 1, frequency 2, frequency 3, total course of treatment: 2 weeks; In the Phase II study, participants will be those with treatment-induced myelosuppression and acute myeloid leukemia/acute lymphoblastic leukemia/primary hematological maligancies who are going to receive hematopoietic stem cell transplantation, UC-MSCs will be preset according to the recommended phase II dose (RP2D) from the Phase Ib study, total course of treatment: 2 weeks.
  Interventions: Biological: umbilical cord derived mesenchymal stem cells

INTERVENTIONS:
Biological: umbilical cord derived mesenchymal stem cells — umbilical cord derived mesenchymal stem cells, intravenous infusion

SUMMARY:
The purpose of the study is to explore the safety and efficacy of umbilical cord derived mesenchymal stem cells in treatment-induced myelosuppression in patients with hematologic malignancies.

DETAILED DESCRIPTION:
Despite the improved prognosis of patients with hematologic malignancies, almost all patients will experience severe myelosuppression induced by anti-cancer treatment, leading to a series of complications such as infection due to neutropenia, bleeding due to thrombocytopenia and/or impaired major organ function such as cardiac function due to anemia, which are the main reasons for dose reduction, dose interrruptions of anti-cancer treatment, failure of hematopoietic stem cell transplantation, and also patients' treatment-related death. It is of significant clinical importance and an urgent need to promote early recovery of myelosuppression and reduce risks of related complications as well as medical burdens. Umbilical cord derived mesenchymal stem cells (UC-MSCs), as a kind of stem cells with multipotential, can widely act on the functional cell units of bone marrow microenvironment and promote the repairment and regeneration of key cells such as hematopoietic stem cells, mesenchymal stem cells and endothelial cells, thus making it an ideal means for effectively promoting recovery of myelosuppression. Patients with hematologic malignancies and treatment-induced myelosuppression will be invited to participate in the Phase Ib/II study, to receive UC-MSCs intravenous infusion and follow-up visits of up to 2 years after enrollment.

ELIGIBILITY:
Inclusion Criteria:

1. Aged between 18 and 75 years old;
2. Either type of primary hematologic malignancies listed below:

   1. Acute myeloid leukemia (AML, AML subtype M3 excluded) or acute lymphoblastic leukemia (ALL) diagosed according to the 2016 revision to the World Health Organization classification of myeloid neoplasms and acute leukemia, either treatment naive participants who are going to receive first induction therapy, or participants who failed first induction therapy and are going to receive re-inducton therapy;
   2. AML or ALL participants who achieved remission and are going to receive consolidation therapy;
   3. Relapsed/refractory AML or ALL participants who are going to receive first re-induction therapy;
   4. Phase II trial will also include: participants with primary hematological maligancies who are going to receive autologous hematopoietic stem cell transplantation (allo-HSCT) whereas are poor mobilizers (CD34+cell count in peripheral blood was below 11-19/μL before collection, or the amount of CD34+ cells transfused was below 2×10^6/kg in allo-HSCT), and the participants' peripheral superficial veins have smooth blood flow which can meet the demand for intravenous drip;
3. The participant or his/her legal guardian is adequately informed of the nature and risks of the study, voluntarily participates in the study with signed informed consent;
4. Male or female;
5. Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0 to 2 (by the day anti-cancer therapy is initiated)
6. Estimated survival of at least 3 months;
7. Adequate major organ function:

   1. Respiratory function: indoor oxygen saturation of at least 95%;
   2. Cardiac function: ejection fraction of left ventricular of at least 45%;
   3. Hepatic function: alanine aminotransferase/aspartate aminotransferase of at most 2.5 times/upper limit of normal value and serum total bilirubin of at most 1.5 times/upper limit of normal value;
   4. Renal function: Serum creatinine of at most 1.5 times/upper limit of normal value;
8. Participants who do not receive any type of anti-cancer therapy within 2 weeks before enrollment (radiation therapy, chemotherapy and/or immune therapy, et al.), and treatment-associated toxicities induced by previous therapy has recovered to Grade 1 or below (except for low grade toxities such as alopecia).

Exclusion Criteria:

1. Overt central nervous system manifestations of hematologic malignancies at diagnosis;
2. Secondary hematological maligancies;
3. Body mass index (BMI) of more than 30 kg/m^2;
4. Myelosuppression induced by conditions other than anti-cancer therapy;
5. Previous radiation therapy performed on sternum or pelvis;
6. Specifically diagnosed and uncontrolled infection at enrollment (Uncontrolled is defined as exhibiting ongoing signs and symptoms of infection without improvement despite anti-infective agents) ;
7. Uncontrolled active bleeding at enrollment;
8. Severe underlying comorbidities affecting survival, including cachexia, severe malnutrition, etc;
9. Estimated survival of at most 48 hours;
10. Active hepatitis B virus (HBV) or hepatitis C virus (HCV) infection;
11. History of or current human immunodeficiency virus (HIV) infection;
12. Continuous usage of immunosuppressants or received organ transplantation in the last 6 months;
13. Participation in clinical trials of other drugs within 6 weeks before enrollment;
14. Previous participation in clinical stem cell research;
15. Receiving any agent concurrently with UC-MSCs infusion which inhibits cell division (hydroxyurea, low-dose cytarabine or methotrexate, etc) ;
16. Severe allergic constitution, or known or suspected allergy to the study drug and its components;
17. Known contraindication to receiving hematopoietic growth factors, transfusion of blood components, anti-infective agents;
18. Female participants who are pregnant or breast feeding;
19. Participants with fertility plan;

    Note: For female participants, they should be surgical sterilized or post-menopausal, or agree to utilize a medically recognised method of contraception (such as intrauterine device, condom) during treatment period of the study and within 6 months after the end of treatment period of the study; For male participants, they should be surgical sterilized or agree to utilize a medically recognised method of contraception (such as intrauterine device, condom) during treatment period of the study and within 6 months after the end of treatment period of the study;
20. Participants suffering from mental illness;
21. Presence of drug abuse/addiction;
22. History of other malignancies other than hematological malignancies within 3 years;
23. Participants without signed informed consent;
24. Participants with poor compliance and are unable to complete the whole course of the study;
25. Participants with circumstances that, in the opinion of the investigator, may increase the risk of the participants or interfere with conduct of the clinical trial and the judgment of results (excessive tension, sensitivity or cognitive impairment, etc) ;
26. Participants with other circumstances that are ineligible for enrollment in this study, in the opinion of the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 181 (Estimated)
Dates: Start 2023-01-01 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2025-01-31 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicities（DLT) | 4 days after the last UC-MSCs dose, up to 12 days
  During the DLT observation period, the subject has an adverse event that is reasonably related to UC-MSCs infusion (possibly, likely or definitely related).
Incidence of Adverse Events (AEs) and Serious Adverse Events (SAEs) | From the day that the last UC-MSCs dose is used to up to 21 days
  To investigate the safety characteristics, percentages will be calculated and grade will be evaluated.
Maximum tolerated dose (MTD) | From the day that the last UC-MSCs dose is used to up to 4 days
  During the dose-escalation phase, the highest dose of dose-limiting toxicity for subjects less than or equal to 1/3 in the dose group of at least 6 evaluble subjects of the study drug after the last UC-MSCs dose.

SECONDARY OUTCOMES:
Time to absolute neutrophil count recovery | From the start of anti-cancer therapy or completion of hematopoietic stem cell transplantation to up to 42 days
  To investigate the efficacy characteristics, time will be measured in days.
Incidence of febrile neutropenia | From the start of anti-cancer therapy or completion of hematopoietic stem cell transplantation to up to 42 days
  To investigate the efficacy characteristics, percentages will be calculated.
Duration of febrile neutropenia | From the start of anti-cancer therapy or completion of hematopoietic stem cell transplantation to up to 42 days
  To investigate the efficacy characteristics, the duration will be measured in days.
Incidence of severe thrombocytopenia | From the start of anti-cancer therapy or completion of hematopoietic stem cell transplantation to up to 42 days
  To investigate the efficacy characteristics, percentages will be calculated.
Time to severe thrombocytopenia recovery | From the start of anti-cancer therapy or completion of hematopoietic stem cell transplantation to up to 42 days
  To investigate the efficacy characteristics, time will be measured in days.
Incidence of severe anemia | From the start of anti-cancer therapy or completion of hematopoietic stem cell transplantation to up to 42 days
  To investigate the efficacy characteristics, percentages will be calculated.
Time to severe anemia recovery | From the start of anti-cancer therapy or completion of hematopoietic stem cell transplantation to up to 42 days
  To investigate the efficacy characteristics, time will be measured in days.
Incidence of infetion | From the start of anti-cancer therapy or completion of hematopoietic stem cell transplantation to up to 42 days
  To investigate the efficacy characteristics, percentages will be calculated.
Duration of infetion | From the start of anti-cancer therapy or completion of hematopoietic stem cell transplantation to up to 42 days
  To investigate the efficacy characteristics, the duration will be measured in days.
Incidence of bleeding | From the start of anti-cancer therapy or completion of hematopoietic stem cell transplantation to up to 42 days
  To investigate the efficacy characteristics, percentages will be calculated.
Duration of bleeding | From the start of anti-cancer therapy or completion of hematopoietic stem cell transplantation to up to 42 days
  To investigate the efficacy characteristics, the duration will be measured in days.
Application rate of blood transfusion | From the start of anti-cancer therapy or completion of hematopoietic stem cell transplantation to up to 42 days
  To investigate the efficacy characteristics, percentages will be calculated.
Application rate of anti-infective agents | From the start of anti-cancer therapy or completion of hematopoietic stem cell transplantation to up to 42 days
  To investigate the efficacy characteristics, percentages will be calculated.
Time to achievement of complete remission | From enrollment to up to 28 days
  To investigate the efficacy characteristics, time will be measured in days.
Duration of complete remission | From enrollment to maximun up to 2 years
  To investigate the safety characteristics, the duration will be measured in days or months.
Event free survival | From enrollment to maximun up to 2 years
  From enrollment to the day of any event.
Overall survival | From enrollment to maximun up to 2 years
  From enrollment to the day of death caused by any reason.
Incidence of infusion reactions in 2 years | 2 years since the last UC-MSCs infusion
  To investigate the safety characteristics, percentages will be calculated.
Incidence of secondary tumor in 2 years | 2 years since the last UC-MSCs infusion
  To investigate the safety characteristics, percentages will be calculated.
Cumulative incidence of relapse of primary disease in 2 years | 2 years since the last UC-MSCs infusion
  To investigate the safety characteristics, percentages will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Qiubai Li, Professor, Study Director — Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Locations (3):
- China (3):
  - Wuhan Central Hospital, Wuhan, Hubei
  - Wuhan Union Hospital, Wuhan, Hubei
  - Wuhan Tongji Hospital, Wuhan, Hubei

IPD SHARING:
Plan to Share IPD: No